CLINICAL TRIAL: NCT05988372
Title: Surufatinib and Serplulimab Combined With AG Regimen Compare With AG Regimen as Conversion Therapy for Patients With Locally Advanced Pancreatic Cancer : a Phase II Randomized Controlled PILOT Study (SAGE)
Brief Title: Surufatinib and Serplulimab Combined With AG Regimen Compare With AG Regimen as Conversion Therapy for Patients With Locally Advanced Pancreatic Cancer (SAGE)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming Kuang, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LAPC2023
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Locally Advanced Pancreatic Cancer
Keywords: Locally Advanced Pancreatic Cancer; Conversion Therapy
MeSH Terms: interventions — surufatinib; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surufatinib + Serplulimab+Albumin-paclitaxel + Gemcitabine (Experimental): enrolled, eligible patients receive Surufatinib, Serplulimab, Gemcitabine and Albumin-paclitaxel
  Interventions: Drug: Surufatinib + Serplulimab+Albumin-paclitaxel + Gemcitabine
- Albumin-paclitaxel + Gemcitabine (Experimental): enrolled, eligible patients receive Gemcitabine and Albumin-paclitaxel
  Interventions: Drug: Albumin-paclitaxel + Gemcitabine

INTERVENTIONS:
Drug: Surufatinib + Serplulimab+Albumin-paclitaxel + Gemcitabine — Surufatinib:250mg orally once a day for 3 weeks(3 weeks 1 cycle) Serplulimab:4.5mg/Kg by intravenous infusions on day1 every 3 weeks Albumin-paclitaxel:125mg/m2 by intravenous infusions on day1 and 8 every 3 weeks Gemcitabine:1000mg/m2 by intravenous infusions on day1 and 8 every 3 weeks
  Arms: Surufatinib + Serplulimab+Albumin-paclitaxel + Gemcitabine
Drug: Albumin-paclitaxel + Gemcitabine — Albumin-paclitaxel:125mg/m2 by intravenous infusions on day1 and 8 every 3 weeks Gemcitabine:1000mg/m2 by intravenous infusions on day1 and 8 every 3 weeks
  Arms: Albumin-paclitaxel + Gemcitabine

SUMMARY:
This is a Phase II Randomized Controlled PILOT clinical study. The purpose of this study is to explore the efficacy and safety of surufatinib and serplulimab in combination with albumin-paclitaxel and gemcitabine in the conversion therapy for patients with unresectable locally advanced pancreatic cancer. Furthermore, it compares the efficacy of surufatinib and serplulimab in combination with albumin-paclitaxel and gemcitabine to the albumin-paclitaxel and gemcitabine regimen in the conversion therapy for patients with unresectable locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
A total of 50 participants are expected to be enrolled in this study; 25 will receive the surufatinib and serplulimab in conjunction with albumin-paclitaxel and gemcitabine regimen and 25 will receive the AG regimen. The participants who have been enrolled will initially undergo two cycles of albumin-paclitaxel and gemcitabine induction chemotherapy. The researcher will assess the patients' efficacy based on their imaging results after the second cycle. Patients with PD will be excluded from this trial, and patients with SD, PR, or CR will be enrolled. Patients will be randomly chosen to receive either the AG regimen for 2-4 cycles or the surufatinib combined with serplulimab and AG regimen for 2-4 cycles. Every two cycles, the researcher assessed the effectiveness of the patients' treatments and the potential for R0 resection. Then, patients with PD were removed from the group, those who could be operated were enrolled for surgical resection, and those without PD and unable to undergo surgery were finished with a total of 6 cycles of either the AG regimen chemotherapy or surufatinib combined with serplulimab and the AG regimen chemotherapy. Within 12 weeks of surgery, patients underwent 0-2 cycles of chemotherapy with the AG regimen or surufatinib combined with serplulimab and AG regimen, totaling 6 cycles of postoperative chemotherapy. Then patients of AG group will enter follow up stage. Patients with R0 resection will accept surufatinib in combination with serplulimab maintenance for no longer than 12 cycles after surgery, or until intolerability, progressive disease, death, or other criteria for study treatment discontinuation specified in the protocol, whichever comes first. Patients who have not progressed and are unable to undergo surgery, or who accepted R1 or R2 resection, after six cycles of the surufatinib combination with serplulimab and AG regimen, will receive sulfatinib combined with serplulimab maintenance therapy for a maximum of 29 cycles, or until intolerance, disease progression, death, or other criteria specified in the study protocol were met.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the patient prior to treatment.
2. Pathologically confirmed unresectable locally advanced pancreatic cancer, received no surgical therapy.
3. Age between 18 and 75 years at the time of study entry.
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
5. Measurable or evaluable lesions according to RECIST v1.1 criteria.
6. Life expectancy ≥ 12 weeks.
7. There are no serious organic diseases of the heart, lungs, brain and other organs.
8. Adequate functioning of the bone marrow and major organs function meeting the following criteria:

   1. White blood cell count ≥ 4 × 109/L, Neutrophil count ≥ 1.5 × 109/L, Platelets count ≥ 100 × 109/L,Hemoglobin ≥ 90 g/L.
   2. Normal coagulation function, without active bleeding or thrombotic diseases: INR ≤ 1.5 × ULN, APTT ≤ 1.5 × ULN.
   3. Liver function: Total serum bilirubin ≤ 1.5 ×ULN, Serum aspartate aminotransferase (AST) and serum alanine aminotransferase (ALT) ≤ 3 × ULN, Obstructive Jaundice with total serum bilirub ≤ 1.5 x ULN after internal/ external drainage.
   4. Kidney function: Serum creatinine ≤ 1.5 × upper limit of normal (ULN) or creatinine clearance ≥ 60 mL/min.
   5. Cardiac function:left ventricular ejection fraction (LVEF) of 50%≥ on 2D cardiac ultrasound.
9. Male or female patients of potential for childbearing who voluntarily used effective contraceptive methods such as double-barrier contraception, condoms, oral or injection avoidance or pregnancy medications, IUDs, etc during the study period and within 6 months of the last study medication . All female patients will be considered fertile unless the female patient is naturally menopausal.

Exclusion Criteria:

1. Participants diagnosed pancreatic cancer with distant metastases.
2. Participation in other antineoplastic drug clinical trials within 4 weeks prior to enrollment;
3. Previous systemic antitumor therapy (chemotherapy, radiation, targeted or immunoth, etc.).
4. Diagnosis of any second malignancy, except for adequately treated basal cell skin cancer or in situ carcinoma of the cervix uteri.
5. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
6. Active or prior documented autoimmune or inflammatory disorders.
7. Participants are being treated with immunosuppressants, or systemic or absorbable topical hormones for immunosuppressive purposes (dose> 10 mg/day prednisone or other equivalent hormones) , and the use is still continued within 2 weeks before enrollment.
8. Have undergone any surgery (other than biopsy) or invasive treatment or manipulation within 4 weeks prior to enrollment and the surgical incision has not healed completely (except intravenous catheterization, puncture drainage, internal or external drainage of obstructive jaundice, etc.)
9. Participants with abnormal thyroid function who were unable to maintain thyroid function within the normal range with medical treatment.
10. Hypertension that cannot be controlled in the presence of optimal treatment is defined as systolic blood pressure ≥ 150 mmHg and/or diastolic blood pressure ≥ 100 mmHg.
11. Urinary routine showed that urinary protein ≥2+, and 24-hour urinary protein>1.0g.
12. Participantst currently has any disease or condition that affects the absorption of the drug, or the participants cannot take sulfatinib orally
13. participants with evidence or history of significant bleeding tendency within 3 months prior to enrollment (bleeding>30 mL within 3 months with hematemesis, melena, hematochezia), hemoptysis (fresh blood>5 mL within 4 weeks); Patients with history of hereditary or acquired bleeding or coagulation dysfunction, with clinically significant bleeding symptoms or definite bleeding tendency within 3 months, such as gastrointestinal bleeding and hemorrhagic gastric ulcer.
14. Cardiovascular disease of significant clinical significance, including but not limited to acute myocardial infarction, severe/unstable angina, or coronary bypass grafting within 6 months prior to enrollment; New York Heart Association (NYHA) grade > 2 for congestive heart failure; ventricular arrhythmias requiring drug therapy; Electrocardiogram (ECG) showing QT interval ≥480 ms;
15. Severe infection that is active or uncontrolled:

    1. Inherited or acquired immunodeficiency disease,
    2. Known clinically significant history of liver disease, including viral hepatitis [known hepatitis B virus (HBV) carriers must exclude active HBV infection , HBV DNA positive (>1×104 copies/mL or >2000 IU/ml)];
    3. known hepatitis C virus infection (HCV) and positive HCV RNA (>1×103 copies/ml) or other hepatitis, cirrhosis.
16. Pregnant or lactating women or participants with family planning during the trial period.
17. Participants have a known history of psychotropic substance abuse, alcoholism, or drug abuse.
18. The investigator believes that the participant has any clinical or laboratory abnormalities or other reasons that are unsuitable for this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-23 (Estimated); Primary Completion 2023-10-23 (Estimated); Study Completion 2026-10-23 (Estimated)

PRIMARY OUTCOMES:
R0 Surgical Resection Rate | Up to 2 years
  Proportion of patients with negative microscopic margins (no tumor cell remains)

SECONDARY OUTCOMES:
Surgical conversion rate | Up to 2 years
  Surgical conversion rate: the proportion of patients with successful conversion and surgical resection in all patients, surgical conversion rate =(number of patients with successful conversion and surgical resection/total number of patients) ×100%.
Objective response rate (ORR) | Up to 2 years
  ORR is defined as the percentage of patients who have achieved complete response (CR) or partial response (PR), as measured by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
Deepness of response (DpR) | Up to 2 years
  DpR is defined as the percentage of maximal tumor reduction from baseline of a target lesion.
Progression-Free Survival (PFS) | Up to 2 years
  PFS is defined as the time from the first dose of administration to progression or death
Disease-free survival (DFS) | Up to 2 years
  DFS is defined as the time interval between the date of enrollment and the date of the first documented evidence of relapse after radical resection at any site or death related to cancer
Over Survival (OS) | Up to 2 years
  OS is defined as the time from first treatment to death, regardless of disease recurrence
Quality of Life (QOL) | Up to 2 years
  Acording the EORTC QLQ-C30.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China